CLINICAL TRIAL: NCT00317902
Title: An Open-Label Study to Evaluate The Effect of Every Other Week PROCRIT (Epoetin Alfa) Dosing (40,000-60,000 Units) On Maintaining Quality of Life and Target Hemoglobin Levels in Anemic HIV-Infected Patients
Brief Title: An Open-Label Study to Evaluate the Effect of Every Other Week PROCRIT� (Epoetin Alfa) Dosing (40,000-60,000 Units) On Maintaining Quality of Life and Target Hemoglobin Levels in Anemic HIV-Infected Patients (CHAMPS II)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ortho Biotech Products, L.P. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR005131
Record Dates: First submitted 2006-04-21; First posted 2006-04-25 (Estimated); Last update posted 2011-05-19 (Estimated); Status verified 2010-04

CONDITIONS: Anemia; HIV Infections
Keywords: Anemia; erythropoetin; Epoetin alfa; erythropoetin recombinant; HIV, AIDS
MeSH Terms: conditions — Anemia; HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Epoetin Alfa

INTERVENTIONS:
Drug: Epoetin alfa

SUMMARY:
The objective of this study was to treat anemic (Hemoglobin (Hb) < 12 g/dL) HIV-infected subjects with once weekly (QW) PROCRIT (Epoetin alfa) to a target Hb of > 13 g/dL and then to assess if the target Hb level and improvements in Quality of Life (QOL) could be maintained with every other week (Q2W) PROCRIT (Epoetin alfa) dosing.

DETAILED DESCRIPTION:
This was a Phase IV, open-label, non-randomized, multi-center study conducted in community based practices, physicians networks, or academic institutions in the US. This study included anemic (Hb < 12 g/dL) HIV-infected subjects and HIV/hepatitis C (HCV) co-infected subjects not receiving HCV treatment on a stable anti-retroviral therapy (ART) regimen for at least 4 weeks prior to enrollment.

Quality of life assessments, laboratory results, and transfusion information were obtained during the study. Laboratory tests, vital signs (blood pressure), and incidence and severity of adverse events were collected and assessed.

The primary objective of this study was to assess if every other week PROCRIT (Epoetin alfa) dosing can maintain quality of life in anemic HIV-infected patients. The primary hypothesis of interest was that the mean quality of life score (as measured by MOS-HIV General Health Perception score) at the end of the every other week (Q2W) maintenance phase was not lower than that at the beginning of the maintenance phase by more than 7 points.

It was anticipated that less frequent dosing, every other week, was more convenient for patients and will improve patient compliance. The starting dose (Baseline/Study Day 1) of PROCRIT (Epoetin alfa) for all eligible subjects was 40,000 U given subcutaneously QW. The maximum duration was 24 weeks. Subjects who achieved target Hb levels >= 13 g/dL were converted to a maintenance dose of PROCRIT (Epoetin alfa) sc Q2W.

ELIGIBILITY:
Inclusion Criteria:

* Understand and sign written informed consent
* HIV-infected patients (as documented by HIV-RNA values)
* HIV/HCV co-infected patients not receiving treatment
* Hemoglobin < 12 g/dL unrelated to transfusion
* Estimated life expectancy of > 9 months
* Has been maintained on a stable antiretroviral regimen for at least four weeks prior to enrollment into this study.

Exclusion Criteria:

* Acute, symptomatic opportunistic infection or other acute AIDS defining illness
* Anemia attributable to factors other than HIV infection (i.e., iron, B12 or folate deficiencies, hemolysis, gastrointestinal bleeding)
* HCV co-infected patients who are anticipated to receive treatment with ribavirin/interferon during the study period. Previous treatment with ribavirin/interferon must have been completed at least 12 weeks prior to study entry
* Ferritin level < 40 ng/mL
* Uncontrolled or severe cardiovascular disease including recent (< 6 months) myocardial infarction, uncontrolled hypertension or congestive heart failure

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 292 (Actual)
Dates: Start 2002-10; Study Completion 2004-05 (Actual)

PRIMARY OUTCOMES:
The primary objective of this study was to assess if every other week PROCRIT (Epoetin alfa) dosing can maintain quality of life (QOL) in anemic HIV-infected patients between Week 24 (or the last measurement) and the beginning of the maintenance phase

SECONDARY OUTCOMES:
The effect of every other week PROCRIT (Epoetin alfa) dosing on maintaining target hemoglobin levels (>13 g/dL), transfusion utilization and safety in anemic HIV-infected patients measured from the beginning of the maintenance phase to Week 24.

CONTACTS AND LOCATIONS:
Overall Officials: Ortho Biotech Products, L.P. Clinical Trial, Study Director — Ortho Biotech Products, L.P.

REFERENCES:
- [Derived] Levine AM, Salvato P, Leitz GJ; Champs 2 Study Group. Efficacy of epoetin alfa administered every 2 weeks to maintain hemoglobin and quality of life in anemic HIV-infected patients. AIDS Res Hum Retroviruses. 2008 Feb;24(2):131-9. doi: 10.1089/aid.2006.0200. PMID 18284320
- See also: An Open-Labeled Study to Evaluate The Effect of Every Other Week PROCRIT (Epoetin alfa) Dosing on Maintaining Quality of Life and Target Hemoglobin Levels in Anemic HIV-Infected Patients — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=931&filename=CR005131_CSR.pdf